CLINICAL TRIAL: NCT05254262
Title: An Observational Multicenter National Trial of Clinical Results and Morbimortality of Surgical Elderly Patients
Brief Title: Multicenter National Trial of Clinical Results of Surgical Elderly Patients
Acronym: CiruGerES:
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, David Parés MD, PhD, Professor of Surgery and Principal Investigator, Germans Trias i Pujol Hospital
Other Study IDs: CiruGerES-1
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-02

CONDITIONS: Surgery--Complications; Age Problem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly patients: Patients age 70 or older, who are admitted in hospital for surgical operation (elective or emergency surgery)
  Interventions: Procedure: Elderly surgical patients

INTERVENTIONS:
Procedure: Elderly surgical patients — Patients who needs elective or emergency surgery for any reason

SUMMARY:
The aim of this study is to study clinical results including mrobidity and mortality of elderly patients (age > 75 years) in Spain during a 3-month period.

DETAILED DESCRIPTION:
The aim of the study it is to analyze the morbidity and mortality of patients older tha 70 admitted on hospital and who needs surgical operation. The results will be analysed in relationship with surgical risk calculator in order to know if it would be posssible to predict morbi-mortality of these cohort of patirents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an age of 70 years old or older
* Admitted on hospital (minimum 1 day of hospital length)
* Needing surgery

Exclusion Criteria:

* Day case -surgery

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with and age of 70 years old or older
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 day
  Patients death during hospitalization or first 30 days after surgery
Complications | 30 day
  Any complication during admission or 30 day after

SECONDARY OUTCOMES:
ASA score | preoperative
  Assessment of surgical risk
ACS NSQIP surgical risk score | preoperative
  Assessment of surgical risk

CONTACTS AND LOCATIONS:
Overall Officials: David Parés, MD, PhD, Principal Investigator — Department of Surgery, Hospital Germans Trias i Pujol
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No